CLINICAL TRIAL: NCT06116526
Title: Dupilumab De-escalation in Pediatric Atopic Dermatitis: A Pilot Trial
Brief Title: Dupilumab De-escalation in Pediatric Atopic Dermatitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00405441
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants are unblinded to the trial arm. Clinical outcomes will be assessed by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dupilumab - discontinuation (Experimental): Participants will discontinue their dupilumab treatment for atopic dermatitis.
  Interventions: Drug: Dupilumab - Discontinuation
- Dupilumab - dose reduction (Experimental): Participants whose standard dupilumab dosing for atopic dermatitis is 200 mg or 300 mg every 2 weeks will decrease drug administration to every 4 weeks, and participants whose standard dupilumab dosing is 200 mg or 300 mg every 4 weeks will decrease administration to every 8 weeks.
  Interventions: Drug: Dupilumab - Dose Reduction
- Dupilumab - standard dosing (Experimental): Participants will continue to receive standard maintenance dupilumab dosing for atopic dermatitis according to FDA labeling, as indicated below.
  Infants ≥6 months and Children <6 years:
  5 to <15 kg: 200 mg every 4 weeks. 15 to <30 kg: 300 mg every 4 weeks
  Children ≥6 years and Adolescents ≤17 years:
  15 to <30 kg: 300 mg every 4 weeks 30 to <60 kg: 200 mg every other week
  ≥60 kg: 300 mg every other week
  Interventions: Drug: Dupilumab - Standard Dose

INTERVENTIONS:
Drug: Dupilumab - Discontinuation — Drug injections are discontinued.
  Other Names: Dupixent
  Arms: Dupilumab - discontinuation
Drug: Dupilumab - Dose Reduction — The drug is given as a subcutaneous injection.
  Other Names: Dupixent
  Arms: Dupilumab - dose reduction
Drug: Dupilumab - Standard Dose — The drug is given as a subcutaneous injection.
  Other Names: Dupixent
  Arms: Dupilumab - standard dosing

SUMMARY:
This is a pilot investigator-blinded, randomized clinical trial to assess the feasibility of dupilumab treatment discontinuation or dose-reduction in children aged 1-17 years who have achieved sustained atopic dermatitis (AD) control on dupilumab.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of three groups: discontinuation of dupilumab; reduction of dupilumab dose; or continuation of standard dupilumab dose. During the active study treatment period, participants will be asked to complete 5 study visits. At these visits, a physician will conduct a skin examination to assess atopic dermatitis (AD) severity and participants will complete questionnaires about their AD symptoms and severity. During the observational period, participants will be asked to complete questionnaires about their AD symptoms and medication use every twelve weeks, for a total of 3 follow-up contacts. The purpose of this study is to evaluate the feasibility and sustainability of reducing or discontinuing dupilumab in children with well-controlled AD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 to <18 years old, either sex, any race or ethnicity
* Provide signed informed consent by parent or legal guardian and informed assent if applicable
* Has a physician confirmed diagnosis of atopic dermatitis
* Has received dupilumab for at least 12 months for the treatment of atopic dermatitis
* Has had well-controlled atopic dermatitis on dupilumab within last 6 months (defined as POEM<=7, EASI<=7, or IGA<=2)
* Able to speak English
* Able and willing to adhere to all study procedures

Exclusion Criteria:

* Taking concurrent systemic medication for atopic dermatitis (e.g., methotrexate, cyclosporine, tralokinumab, abrocitinib, upadacitinib, systemic corticosteroids)
* Using concurrent phototherapy for atopic dermatitis
* Taking dupilumab for a clinical indication other than atopic dermatitis (such as asthma or eosinophilic esophagitis)
* Poor control of atopic dermatitis
* Poor control of asthma or eosinophilic esophagitis
* Has used an investigational drug within 90 days or plan to use an investigational drug during the study period
* Does not have health insurance or will lose health insurance during the study period

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Successful Dose Reduction of Dupilumab | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  Successful de-escalation is defined as maintaining a reduced dose (i.e., less frequent administration) of dupilumab after initial de-escalation on week 0. Patients who require re-escalating the dose of dupilumab to standard dosing or adding other systemic treatments for their AD will be regarded as treatment failure.
Percentage of Participants with Successful Discontinuation of Dupilumab | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  Successful discontinuation is defined as maintaining discontinuation of dupilumab after initial discontinuation on week 0. Patients who require resumption of dupilumab or beginning other systemic treatments for their AD will be regarded as treatment failure.

SECONDARY OUTCOMES:
Change in Investigator's Global Assessment (IGA) Scores | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  IGA is a global clinical assessment scale to determine severity of AD and clinical response to treatment on a static 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on the degree of erythema and papulation/infiltration. The IGA score ranges from 0 to 4. Higher scores indicate greater severity of AD.
Change in Eczema Area and Severity Index (EASI) Scores | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The EASI score is used to evaluate severity of AD based on AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. The total EASI score ranges from 0 to 72. Higher scores indicate greater severity of AD.
Change in Patient Oriented Eczema Measure (POEM) Scores | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The POEM is a 7-item questionnaire to assess disease symptoms in children and adults with AD. It is composed of 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) based on symptom frequency during the past week (0 = 'no days', 1 = '1 to 2 days', 2 = '3 to 4 days', 3 = '5 to 6' days, and 4 = 'every day'). The total POEM score ranges from 0 to 28. Higher scores indicate more severe disease and poor quality of life.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Itch questionnaire score | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The PROMIS Itch questionnaire measures the extent to which patients experience problems with itchiness over the past 7 days using a 5-point Likert scale (1 = Never; 2 = Rarely; 3 = Sometimes; 4 = Often; and 5 = Almost Always). Higher scores reflect greater severity of experienced itch symptoms.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Problem questionnaire score | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The PROMIS Sleep Problem questionnaire measures the extent to which patients experience problems with sleep over the past 7 days using a 5-point Likert scale (1 = Never; 2 = Almost never; 3 = Sometimes; 4 = Almost always; and 5 = Always). The sleep problems contain sleep disturbances (sleep quality, sleep onset, sleep continuity) and sleep-related impairment (perceptions of sleepiness during usual awake hours and reported impairments during the day associated with sleep problems or daytime sleepiness). Higher scores reflect greater severity of sleep problems.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety questionnaire score | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The PROMIS Anxiety questionnaire measures the extent to which patients experience problems with anxiety over the past 7 days using a 5-point Likert scale (1 = Never; 2 = Almost never; 3 = Sometimes; 4 = Often; and 5 = Almost Always). The questionnaire includes fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), social/separation anxiety (fear or distress when separating from caregivers), and somatic symptoms related to arousal (racing heart, dizziness). Higher scores reflect greater severity of experienced anxiety symptoms.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depressive Symptoms questionnaire score | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The PROMIS Depressive Symptoms questionnaire measures the extent to which patients experience problems with depression over the past 7 days using a 5-point Likert scale (1 = Never; 2 = Almost never; 3 = Sometimes; 4 = Almost Always; and 5 = Always). The depressive symptoms include negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation); decreased positive affect, anhedonia (loss of interest, inability to engage in play), and engagement. Higher scores reflect greater severity of experienced depressive symptoms.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function questionnaire score | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The PROMIS Cognitive Function questionnaire measures the extent to which patients experience problems with cognitive function over the past 4 weeks using a 5-point Likert scale (1 = All of the time; 2 = Most of the time; 3 = Some of the time; 4 = A little of the time; and 5 = None of the time). The questionnaire includes difficulties in cognitive abilities (e.g., memory, attention, and decision making), and difficulties in the application of such abilities to everyday tasks (e.g., planning, organizing, calculating, remembering, and learning). Lower scores reflect greater impact on cognitive function.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health questionnaire score | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The PROMIS Global Health questionnaire measures the extent to which patients experience problems with global health in general using a 5-point Likert scale (1 = Poor; 2 = Fair; 3 = Good; 4 = Fair; and 5 = Excellent). The questionnaire includes an overall evaluation of physical, mental health, and social health. Higher scores reflect a lower quality of global health.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity questionnaire score | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The PROMIS Pain Intensity questionnaire measures the intensity of patients' pain due to their AD over the past 7 days using a 10 point scale, with 0 indicating "No Pain" and 10 indicating "the worst pain possible." Higher raw scores reflect greater severity of experienced pain due to AD.
Change in Children's Dermatology Life Quality Index (CDLQI) score | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  CDLQI is a 10-item questionnaire to assess the impact of skin problems on the quality of life of children between the ages of 4-16 years old over the last one week. Each question is evaluated on a 4-point scale: Not at all = 0, A Little = 1, Quite A Lot = 2, Very Much = 3. Higher scores indicate worse child-reported quality of life. CDLQI scores indicate the degree of severity burden on the quality of life: No effect = 0-1; Small effect = 2-6; Moderate effect = 7-12; Very large effect = 13-18; and Extremely large effect = 19-30.
Change in Family Dermatology Life Quality Index (FDLQI) score | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  FDLQI is a 10-item questionnaire to assess the impact of skin problems on the quality of life of families over the last one month. Each question is evaluated on a 4-point scale: Not at all = 0, A Little = 1, Quite A Lot = 2, Very Much = 3. Higher scores indicate worse quality of life. FDLQI scores indicate the degree of severity burden on the quality of life: No effect = 0-1; Small effect = 2-6; Moderate effect = 7-12; Very large effect = 13-18; and Extremely large effect = 19-30.
Changes in Utilization of Topical Medications for Atopic Dermatitis | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  Participants will provide a self-report of their daily utilization of topical medications (medication name, dose and frequency) using a paper-form Daily Diary.
Adverse Events After Dupilumab Dose-reduction or Discontinuation | From Baseline through Week 16 (active protocol phase) and Week 17 through Week 52 (observational phase)
  The number of participants who experience adverse events ≥ Grade 2 is based on the Common Terminology Criteria for Adverse Events (CTCAE). The CTCAE is generally graded as follows: Grade 1 - mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not needed; Grade 2 - moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living; Grade 3 - severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limited self care activities of daily living; Grade 4 - life-threatening consequences; urgent intervention indicated; Grade 5 - death related to adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Joy Wan, MD MSCE, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Univerisity, Baltimore, Maryland, United States

REFERENCES:
- [Background] Drucker AM, Wang AR, Li WQ, Sevetson E, Block JK, Qureshi AA. The Burden of Atopic Dermatitis: Summary of a Report for the National Eczema Association. J Invest Dermatol. 2017 Jan;137(1):26-30. doi: 10.1016/j.jid.2016.07.012. Epub 2016 Sep 8. PMID 27616422
- [Background] Langan SM, Irvine AD, Weidinger S. Atopic dermatitis. Lancet. 2020 Aug 1;396(10247):345-360. doi: 10.1016/S0140-6736(20)31286-1. PMID 32738956